CLINICAL TRIAL: NCT01632254
Title: Study to Investigate the Sensitivity and Specificity of 3.0 Tesla MRI, MRS and Ultrasound Imaging for Carotid Artery Plaque Dimension and Composition Assessment
Brief Title: Study to Investigate the Sensitivity and Specificity of 3.0 Tesla MRI for Carotid Artery Plaque
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, E.S.stroes, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: TIP-H
Record Dates: First submitted 2011-10-13; First posted 2012-07-02 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-05

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with ≥70% carotid artery stenosis

SUMMARY:
The aim of this study is to develop non-invasive MRI, and MRS approaches that will quantify the plaque composition and lipid content of plaques and will have the potential for repeated in vivo measurements. To investigate sensitivity and specificity of 3.0 Tesla MRI and MRS for dimension and composition assessment of carotid artery plaques, in particularly those plaques with lipid rich necrotic cores. This non-invasive cross-sectional study, compares carotid parameters of in-vivo 3.0 Tesla MRI, MRS and B-mode ultrasound with histology specimens collected at endarterectomy.

DETAILED DESCRIPTION:
Atherosclerosis is a protracted and in fact lifelong progressive disease. Over time, lipids accumulate in the artery wall forming fatty streaks, which eventually can develop into atherosclerotic plaques (1). The later stages of the process, from quiescent atherosclerotic plaque to an active plaque, have a high risk of triggering acute vascular events, such as myocardial infarction and stroke (1).

Much effort has been put in the development of novel drugs aimed to prevent cardiovascular disease. Low Density Lipoprotein cholesterol (LDL-C) lowering drugs, in particularly statins, play a pivotal role. The hypothesis that serum lipid lowering results in decrease of lipid accumulation in the arterial wall and thus atherogenesis, has formed the basis for successful drug developing strategies (1;2).

To draw valid conclusions on determinants of disease and effectiveness of lipid modifying therapeutic intervention, imaging of atherosclerosis can be used as a validated tool to assess efficacy of novel compounds (3;4).

Although imaging arterial wall dimensions by B-mode ultrasound and intra-vascular ultrasound have proven their value, longitudinal data of the effects of cardiovascular drugs on arterial wall and plaque composition, in particular of vulnerable plaques with lipid rich necrotic cores (LRNC), are scarce.

Magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) are non-invasive imaging modalities that can potentially image plaque composition in-vivo in human carotid arteries. MRI image acquisition at various weightings enables visualisation of plaque composition. Calcification, haemorrhage, fibrous cap and lipid rich necrotic cores can readily be distinguished, providing information on plaque vulnerability. MRS gives a spectrum of resonances, affording detection of specific chemical components through their inherent frequency shift relative to water (5). In image guided MRS, an MR image can be utilized to image and localize a plaque. Proton spectra can then be collected from these plaques, such that the specific proton resonances of lipid components in a mobile state, including cholesterol ester (CE), can be identified (6).

ELIGIBILITY:
Inclusion Criteria:

* Patients are to meet the inclusion criteria of the Athero-Express study.
* These patients are eligible to undergo carotid endarterectomy in either the St. Antonius Hospital, Nieuwegein.
* Willing and able to undergo non-invasive MRI, MRS and ultrasound examinations in the Academic Hospital Center, Amsterdam.
* Signed informed consent

Exclusion Criteria:

* Patients not suitable for MRI (e.g. metal in the body, as a result of pacemaker or artificial cardiac valves); claustrophobia; surgery performed in the neck area of the carotid measurements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ≥70% carotid artery stenosis on clinical ultrasound duplex examination, scheduled for endarterectomy in the Athero-Express study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Plaque characteristics as assessed by 3.0 Tesla MRI. | 1 month
  Total plaque volume, plaque calcification volume, plaque haemorrhage volume, lipid rich necrotic core volume, fibrous cap thickness, as assessed by 3.0 Tesla MRI

SECONDARY OUTCOMES:
Water and lipid content of the plaque as assessed by MRS/3.0T MRI | 1 month
  The ratio of the integrated lipid peak versus the unsuppressed water peak (expressed as a percentage), as assessed by MRS.
Plaque composition and size as assessed by histological analysis | 1 month
  Plaque size, morphology and phenotype (presence of collagen, smooth muscle cells, calcifications, macrophages, thrombus and fat), as assessed by histology analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- See also: Related Info — http://www.amc.nl